CLINICAL TRIAL: NCT02092727
Title: The Reducing Disparities in Access to kidNey Transplantation (RaDIANT) Community Study
Acronym: RaDIANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rachel Patzer, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00056381; 1R24MD008077-01 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Kidney Disease
Keywords: Dialysis facilities; African Americans; Racial disparity; Kidney Transplantation; Community-based Participatory Research; Coalition; Georgia
MeSH Terms: conditions — Kidney Diseases | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard of care arm will receive no specific interventions, but will have access to standard educational materials and quality improvement through End Stage Renal Disease Network 6.
- Behavioral Intervention (Experimental): A variety of dialysis facility-level, behavioral interventions will be examined.
  Interventions: Behavioral: Behavioral Interventions for Dialysis Facilities

INTERVENTIONS:
Behavioral: Behavioral Interventions for Dialysis Facilities — 1. Educational seminars and monthly educational webinars
  2. Peer-to-peer mentoring program
  3. Bulletin boards about transplantation
  4. Facility-specific feedback reports detailing transplant referral data for their center compared to state average
  5. Formulate a facility-specific improvement plan to increase transplant referrals.
  6. Requirement to form a Patient and Family Advisory Group to increase outreach about transplant education within the facility.
  7. Monthly monitoring and reporting of patient referrals to ESRD Network
  8. Conduct a patient and family education session about transplantation
  9. Host a movie day to show Living ACTS (About Choices in Transplantation & Sharing) video
  Arms: Behavioral Intervention

SUMMARY:
The Southeastern Kidney Transplant Coalition is an academic-community collaboration between partners in the kidney disease community who share the common goal of eliminating health disparities in access to kidney transplantation among African American End Stage Renal Disease living in Georgia, North Carolina, and South Carolina. Volunteer members of this community-based coalition include patients with kidney disease, dialysis facility staff and providers, transplant centers, quality improvement organizations, and patient advocacy organizations. The burden of kidney disease is highest in the Southeast, and yet the rate of kidney transplantation is the lowest in the nation. Further, the investigators research suggests that racial disparities in access to kidney transplantation are concentrated in the Southeast, where African Americans are less likely to access each step in the transplant process. The long-term goal of the investigators Coalition is to use community- based participatory research approaches to develop, test, and disseminate sustainable, community interventions improve access to transplant for African American patients with kidney disease. The Reducing Disparities in Access to kidNey Transplantation (RaDIANT) community study proposes to use community-based participatory research methods to develop a multilevel intervention to reduce racial disparities in access to kidney transplantation. The long-term impact of this application will be to reduce racial disparities in the kidney disease community.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis facilities within GA were considered for this intervention due to data restrictions. The remaining facilities were selected in a step-wise selection process 1) The presence of a racial disparity in referral or 2) a crude referral risk less than six percent.
* The presence of a racial disparity was based on the crude referral risk difference and the standardized referral risk difference.
* The remaining facilities had a calculated 6-month crude referral risk mean of 0.06 and all facilities with a crude referral risk less than the mean were selected for inclusion.
* The final pool of 134 facilities were randomized to either the intervention or control group using a one to one ratio.

Exclusion:

* Facilities with a 6-month population (from June-December 2012) of less than 13 End Stage Renal Disease patients <70 years of age within a facility were excluded.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Referral for Kidney Transplantation | One Year
  Following a multicomponent intervention at the dialysis facility level, change in referral for kidney transplantation from baseline to follow-up (at one year) will be calculated.

SECONDARY OUTCOMES:
Reduction in Racial Disparity | One Year
  Following a multicomponent intervention at the dialysis facility level, reduction in racial disparity (African American vs. Caucasian) of referral for transplantation (from baseline to one year follow up) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Patzer, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Dialysis Facilities throughout the State of Georgia, ESRD Network 6, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hamoda RE, Gander JC, McPherson LJ, Arriola KJ, Cobb L, Pastan SO, Plantinga L, Browne T, Hartmann E, Mulloy L, Zayas C, Krisher J, Patzer RE. Process evaluation of the RaDIANT community study: a dialysis facility-level intervention to increase referral for kidney transplantation. BMC Nephrol. 2018 Jan 15;19(1):13. doi: 10.1186/s12882-017-0807-z. PMID 29334900
- [Derived] Patzer RE, Gander J, Sauls L, Amamoo MA, Krisher J, Mulloy LL, Gibney E, Browne T, Plantinga L, Pastan SO; Southeastern Kidney Transplant Coalition. The RaDIANT community study protocol: community-based participatory research for reducing disparities in access to kidney transplantation. BMC Nephrol. 2014 Oct 28;15:171. doi: 10.1186/1471-2369-15-171. PMID 25348614